CLINICAL TRIAL: NCT04600882
Title: Characterization of a Clinical Subpopulation in Children With Autism Spectrum Disorder (ASD)
Brief Title: Characterization of a Clinical Subpopulation in Children With Autism Spectrum Disorder
Status: Withdrawn | Type: Observational
Why Stopped: No subjects enrolled
Sponsor: Stalicla SA (Industry)
Responsible Party: Sponsor
Other Study IDs: STP1-C002
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorder; endophenotyping; observational
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This single-center, observational study is being conducted to identify a well-characterized subgroup within the ASD patient population, based on clinical symptoms and biosample analysis.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with ASD (based on DSM-5 criteria and supported by either ADI-R or ADOS-2 scores)
* At least two well documented head circumference values recorded within the first 2 years of life
* Participants must have a parent or reliable caregiver who agrees to provide information about the participant as required by the protocol and should be fluent in English

Exclusion Criteria:

* Genetically identified ASD (syndromic form of autism, e.g. fragile X)
* Episode of fever (i.e. ≥100.5 °F) or clinically significant illness without fever (as judged by the Investigator), within 10 days before the study visit

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Nationwide Children's Hospital Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of non-behavioral phenotypical traits in sub-populations with Autism Spectrum Disorder (ASD) | Day 0
  A questionnaire will be administered to collect non-behavioral traits and co-occurring conditions data of the participants

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States